CLINICAL TRIAL: NCT07300111
Title: A Randomized, Open Label, Active-controlled, Parallel-group, Multi-center Study to Evaluate Efficacy and Safety of QLG1218(Daprodustat) in Chinese Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease.
Brief Title: A Study to Evaluate Efficacy and Safety of QLG1218(Daprodustat) in Chinese Hemodialysis (HD)-Dependent Subjects With Anemia Associated With Chronic Kidney Disease (CKD)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLG1218-301
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Darbepoetin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daprodustat (Experimental)
  Interventions: Drug: Daprodustat
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Daprodustat — Subjects will receive oral daprodustat once daily for 28 weeks
  Arms: Daprodustat
Drug: Darbepoetin alfa — Subjects will receive IV darbepoetin alfa once weekly for 28 weeks
  Arms: Darbepoetin alfa

SUMMARY:
This study is to evaluate the efficacy and safety of QLG1218(daprodustat) following a switch from erythropoiesis-stimulating agent (ESA) in Chinese HD subjects with renal anemia who are currently treated with ESA. The primary objective is to demonstrate non-inferiority of QLG1218 to darbepoetin alfa. This study is a randomized, open Label, active-controlled, parallel-group, multi-center Study. The total duration of the study will be approximately 32 weeks including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male，age 18 to 75
2. Weight 45 to 100 kg
3. Receiving hemodialysis (including hemodiafiltration) consistently three times a week for at least 12 weeks prior to screening.
4. Patients with pre-dialysis Hb levels measured after the maximum interdialytic interval at Scr Visit 1 and Scr Visit 2 (1 week after the start of observation) of ≥95 g/L and <120 g/L and a difference (in absolute value) between Scr Visit 1 and Scr Visit 2 of ≤15 g/L.
5. TSAT >20% and ferritin >100 μg/L
6. Use of one and the same ESA for 10 weeks prior to screening
7. Darbepoetin alfa 10 to 60 μg per week, epoetin (including biosimilars) 1500 to 10000 international units (IU) per week.

Exclusion Criteria:

1. History of bone-marrow hypoplasia, pure red cell aplasia, pernicious anemia, thalassemia, sickle cell anemia, or myelodysplastic syndromes.
2. History of malignancy.
3. Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within 12 weeks prior to screening or during a period from screening to Day 1.
4. Myocardial infarction, acute coronary syndrome, stroke, or transient ischemic attack: Diagnosed within 12 weeks prior to screening or during a period from screening to Day 1
5. Chronic Class III or IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
6. poorly controlled hypertension.
7. Current unstable active liver or biliary disease.
8. History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
9. Use or planned use of any prescription or non-prescription drugs or dietary supplements that are prohibited during the study period.
10. Use of an investigational agent within 30 days or five half lives of the investigational agent (whichever is longer)
11. Use of daprodustat or other HIF-PHI within 4 weeks prior to screening, or any prior treatment with daprodustat for a treatment duration of > 4weeks.
12. QTc >500 milliseconds (msec); or QTc >530 msec in subjects with bundle branch block.
13. ALT or AST >2 upper limit of normal (ULN)，or bilirubin >1.5×ULN.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Mean Hemoglobin (Hgb) During the Efficacy Evaluation Period | Weeks 25 to 28
  The mean hemoglobin during the Evaluation Period was estimated by a statistical model.